CLINICAL TRIAL: NCT04665492
Title: Electroencephalographic Predictors of Central Neuropathic Pain in Subacute Spinal Cord Injury
Brief Title: EEG Predictors of Neuropathic Pain in SCI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Buckinghamshire Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: GN20NE240; 280703 (Other: IRAS)
Record Dates: First submitted 2020-11-16; First posted 2020-12-11 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Central Neuropathic Pain; Spinal Cord Injuries
Keywords: Spinal Cord Injury; Central Neuropathic Pain; EEG; Pain markers
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SCI with CNP: People with subacute spinal cord injury and no chronic pain
  Interventions: Diagnostic Test: EEG recording 1; Diagnostic Test: EEG recording 2; Diagnostic Test: Sensory Test; Diagnostic Test: Brief Pain Inventory 1; Diagnostic Test: Multidimensional health locus of control; Diagnostic Test: Sensory test thermal; Diagnostic Test: Neuropathic pain symptoms; Diagnostic Test: McGill pain questionnaire; Diagnostic Test: Pain Catastrophising Scale
- SCI no CNP: People with subacute spinal cord injury with central neuropathic pain
  Interventions: Diagnostic Test: EEG recording 1; Diagnostic Test: EEG recording 2; Diagnostic Test: Sensory Test; Diagnostic Test: Brief Pain Inventory 1; Diagnostic Test: Sensory test thermal; Diagnostic Test: Neuropathic pain symptoms
- Able bodied: Able bodied people with no chronic pain
  Interventions: Diagnostic Test: EEG recording 1; Diagnostic Test: Brief Pain Inventory 1

INTERVENTIONS:
Diagnostic Test: EEG recording 1 — Multichannel EEG recording in eyes opened and eyes closed relaxed state and during imagined movement (all one experimental session). EEG device "usbamp" (company "Guger Technologies", Austria) will be used.
Diagnostic Test: EEG recording 2 — Multichannel EEG recording in eyes opened and eyes closed relaxed state and during imagined movement (all one experimental session). This intervention will take place six month after EEG recording 1. EEG device "usbamp" (company "Guger Technologies", Austria) will be used.
  Groups: SCI no CNP; SCI with CNP
Diagnostic Test: Sensory Test — Test for mechanical sensations of the feet and shins of both legs as well as on the trapezoidal muscle on both sides. Semmes-Weinstein Monofilaments will be used
  Groups: SCI no CNP; SCI with CNP
Diagnostic Test: Brief Pain Inventory 1 — This questionnaire that ask about any acute or chronic pain
Diagnostic Test: Multidimensional health locus of control — Questionnaire that test personal belief about control of one's own health
  Groups: SCI with CNP
Diagnostic Test: Sensory test thermal — Test of thermal sensations (thermal roller) of the feet and shins of both legs as well as on the trapezoidal muscle on both sides. A "Somedic SenseLab Rolltemp" device will be used
  Groups: SCI no CNP; SCI with CNP
Diagnostic Test: Neuropathic pain symptoms — Questionnaire that test for neuropathic pain symptoms
  Groups: SCI no CNP; SCI with CNP
Diagnostic Test: McGill pain questionnaire — Questionnaire assess three separate components of experiencing pain; the sensory intensity, the emotional impact and the cognitive evaluation of pain.
  Groups: SCI with CNP
Diagnostic Test: Pain Catastrophising Scale — Questionnaire use to identify individual pain experience.
  Groups: SCI with CNP

SUMMARY:
Spinal cord injury (SCI), induced by damage to the spinal cord, can cause life-altering levels of disability including the development of chronic pain. Central Neuropathic Pain (CNP) typically develops within months after injury in 40-50% of SCI patients, affecting everyday activity, sleep and mood. There is no cure for CNP, it can be very difficult to treat and is often refractory to any pharmacological treatments.

In a previous study (study no. 14/WS/1029) the principle investigators showed that the likelihood of CNP developing can be predicted by defining characteristics of brain waves that are related to pain. We will use electroencephalograph (EEG) to measure brain activity in people early after SCI, before they develop pain, knowing that about half will develop pain within a year. We aim to recruit 80 participants, aged 18-80; 40 with subacute spinal injury (level C3-T12) and no symptoms of CNP; 20 with symptoms of CNP and 20 able-bodied participants. Completeness of injury is irrelevant. Patients will be recruited by clinical consultants within national spinal units in Glasgow and Stoke Mandeville. Patients will undergo two EEG recording sessions in which they will imagine movements while we record EEG. Sessions will also involve basic sensory testing and completion of questionnaires. Able-bodied participants will be recruited by the Philosophy Doctor (PhD) candidate at the University of Glasgow and undergo only one EEG session (identical to SCI patients).

The primary aim of this study is to use early EEG markers of CNP to optimise and validate an existing computer program based on machine learning to enable more accurate prediction of pain in newly injured patients with the hope of aiding future treatments. Secondary aims include characterising EEG features which might describe different phases in patients' development of CNP and exploring possible differences between pain at/below the level of SCI based on EEG markers.

DETAILED DESCRIPTION:
Study Design The proposed study will be a longitudinal cohort study in which participants will attend one assessment session as inpatients in the subacute stage and a further assessment six months later, during which time patients are likely to be outpatients. Each session will last up to two hours and questionnaires may be completed within the hospital or outside. To minimise the drop-out, patients will be followed-up though their regular visits to the Queen Elizabeth National Spinal Injuries Uni (QENSIU) or Stoke Mandeville National Spinal Injuries Centre (NSIC) to categorise occurrence of pain, based on the recommended criteria for CNP and the International Spinal Cord Injury Pain Classification System. For those unable to attend the follow-up session, Co-Investigators will take information from their patient notes about their pain, allodynia and hyperalgesia in order to ensure that pain status is collected twice for all participants.

The study will be carried out on 20 able bodied and 60 subacute SCI patients, 40 with no CNP, and 20 with CNP (refer to section 8 for group size considerations). All patients will attend two recording sessions, 2 hours in length, during which time they will undergo EEG recordings as well as sensory testing (including mechanical and thermal tests). This is based on protocol used with the previous cohort. The first test will be carried out as soon as the patients' health condition allows them to sit for the duration of the experiment (this could be within first 3-6 months post injury as Stoke Mandeville Natioanl Spinal Injury Centre (NSIC) does not admit any early injury patients) and the second assessment will take place approximately 6 months later. Able-bodied participants will attend only one session.

Recruitment QENSIU admits around 110 new patients annually whilst Stoke Mandeville Hospital admits around 200. This gives 600 potential volunteers over a 2 year period which should be sufficient to recruit the targeted number. It is planned to recruit approximately half of participants (around 30 people with SCI) from each centre.

Patients will be identified and approached by their clinical consultants (Co-Investigators Dr Mariel Purcell and Dr Maurizio Belci). Prior to participating, patients will be given information sheets and consent forms to sign and should the participant themselves be unable to physically sign, a witnessed proxy can do so on the patient's behalf.

Able bodied participants will be recruited by advertising the study at the University of Glasgow and their data will be collected within the University of Glasgow Rehabilitation Engineering laboratory on University Campus. They will be recruited by the PhD student.

Assessments The patient participants will attend one assessment session as inpatients in the subacute stage and a further assessment six months later. Experimental and data collection procedures will be identical in both the first and second assessments undertaken by patients. This includes EEG recordings, sensory testing and questionnaires. Able bodied participants will only attend one assessment.

Experimental Procedures Questionnaires During assessment sessions, all patients will be asked to complete questionnaires which will allow us collect data on the status of their pain at the time of each visit.

The following questionnaires will be given to patients who at the time of assessment experience CNP:

* Brief Pain Inventory
* McGill pain questionnaire
* Neuropathic Pain Symptoms Inventory
* Multidimensional health locus of control (referring to spinal cord injury as "condition")
* Pain catastrophising scale (referring to the existing pain)

Patients who at the time of first assessment already had pain will be asked to repeat only first two questionnaires on the second assessment, after 6 months. It takes approximately 30 min to fill out all 5 questionnaires. Patients can fill out questionnaires at their own time. Outpatients (second assessment) will receive questionnaires and an envelope with a stamp to post it, or they could alternatively take scan/photos of questionnaires and send them to research team.

Patients with no pain will be asked to complete:

* Brief Pain Inventory
* Multidimensional health locus of control (referring to spinal cord injury as "condition")

Able bodied participants will be asked to fill out the Brief Pain Inventory. All patients with CNP will be diagnosed prior to the study as part of their regular treatment at the hospital. The diagnosis is based on recommendations by the International Spinal Cord Association.

Equipment All equipment has necessary medical device Certificate Europe (CE) mark. Both spinal units (QENSIU and NSIC) and University facilities (for able-bodied assessments) have the same equipment.

Sensory Tests We will use existing clinical American Spinal Injury Association (ASIA) testing information to assess the level and completes of injury i.e. we will gain this information from patient notes following assessment performed by healthcare professional.

All patients will be tested for mechanical and thermal sensations at the foot and shin of both legs and on the trapezoidal muscle on both sides. These are recommended sensory sites from the literature for the following reasons: the feet and shanks are under the level of injury in both tetra and paraplegic patients and are typically reported as locations where most patients with SCI CNP report pain. Trapezoidal muscles are above the level of injury for all patients. Testing only 3 sites on both sides should minimise total assessment time and reduce patients' inconvenience.

Sensory mechanical assessments will comprise a determination of light touch and pinprick which will also serve as a sign of allodynia and hyperalgesia. A mechanical wind up test (with monofilament no. 6.65) will be performed and sensory thermal tests will be conducted using a device named "Rolltemp" (manufacturer "Somedic SenseLab" ). This device consists of two rollers on handles, one roller being warm and the other cold. These are rolled over the skin of the patients who are able to determine the corresponding sensations. Sensory testing will take 30-40 min.

Able bodied participants will not undergo sensory tests.

EEG Recording EEG will be recorded from 64 locations over the entire scalp according to the American Clinical Neurophysiology Society's 10-10 system. EEG will be recorded with a g.Tech biosignal USB amplifier (Guger Technologies, Austria) which enables on-line EEG measurement, signal analysis and visualisation of EEG signals on a computer screen.

Markers of longstanding CNP are present in both spontaneous and induced states such as during motor imagination. As such, EEG activity will first be recorded in the relaxed state of all patients with eyes open and eyes closed (spontaneous EEG), followed by EEG recording during cue-based motor imagination as done previously with the original cohort. This study showed that the presence of CNP affects cortical areas of both paralysed and non-paralysed limbs. Induced EEG will be recorded during cue-based motor imagination where the task will comprise patients sitting in front of a computer screen and undergoing several trials imagining waving their left hand, right hand or tapping both feet. The motor imagery session will be separated into 6 sub sessions each last approximately 5 minutes, to minimise patient discomfort due to tiredness and increased level of concentration. Duration of the EEG recording including setup, breaks and active participation will be up to 1.5 hours. Patients will be allowed to use their mobile phone or to read during the setup period.

In summary, sensory tests and EEG recording will take approximately 2 hours and will be performed on the same day. Filling out self-administered questionnaires will take up to an additional 30 min and may be carried out on the same day or separately. During the first assessment patients will get advice and assistance from researchers when completing the questionnaires. For the second assessment they will be able to fill them out at home on their own.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients with SCI and NO chronic pain are as follows:

* Age between 18-80
* Subacute spinal cord injury (within 6 months post injury)
* Level C3-T12
* ASIA A, B, C or D
* Normal or corrected to normal vision
* No allodynia or hyperalgesia

Inclusion criteria for patients with SCI and CNP are as follows:

* Age between 18-80
* Subacute spinal cord injury (within 6 months of injury)
* Level C3-T12
* ASIA A, B, C or D
* Normal or corrected to normal vision
* Presence of allodynia or hyperalgesia
* Diagnosed CNP related to SCI equal or larger than 4 on visual numerical scale (VNS)

Inclusion criteria for able-bodied participants:

* Age 18-80
* No self-reported neurological conditions
* No chronic or acute pain equal or larger than 3 on VNS
* Normal or corrected to normal vision
* English speaker

Exclusion Criteria:

Exclusion criteria for patients with and without CNP:

* Inability to understand the task
* Inability to sit for at least 2 hours (duration of EEG assessment)
* Invasive 24/7 ventilation
* Previously confirmed brain injury, (peripheral nerve injury and brachial plexus injury)
* Other self-reported neurological condition that would affect EEG recording
* Presence/history of any other chronic or acute pain (larger or equal to 3 on the VNS)
* Pressure sores or any other condition that might prevent sitting for 2 hours
* Halos or neck support that prevent EEG recording
* Infections of the skin or communicable diseases (e.g. hospital bugs)
* Concurrent acute medical problems (e.g. infections)
* Infection control issues i.e. the need for patient isolation
* Do not understand English

Able bodied people and people who had spinal cord injury and are still in subacute phase (6 monthExclusion Criteria for able-bodied participants:

* Unable to give informed consent
* Presence of chronic or acute pain equal to or larger than 3 on VNS
* Any self-reported neurological conditions
* Non-English Speaker s post injury)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Able bodied people and people with subacute spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
EEG based classifier of pain | All groups EEG recording upon recruitment
  Create a software application that can classifify between people with SCI and healthy people and people with SCI with and without pain based on EEG markers
Changes in EEG | EEG recording upon recruitment and EEG recording six month later in all groups of people with SCI
  Difference between baseline EEG and EEG recorded six months later

SECONDARY OUTCOMES:
EEG markers of different phased of SCI | Fist EEG recording upon recruitment, second six month later
  To characterise EEG features which may describe different phases in the development of CNP in SCI which may characterise how EEG markers evolve over time in SCI, starting before the onset of any physical symptoms
EEG markers of at level and below level pain | Fist EEG recording upon recruitment, second six month later
  Anlysis of EEG in people with different types of neuropathic pain (under and at level of injury)
Correlation between sensory and neurological test and questionnaires | Fist EEG recording, sensory test and questionnaires uppon recruitment, second six month later
  To compare and combine EEG predictors using prediction markers evoked in response to peripheral test sensory stimuli (e.g. mechanical, thermal stimuli)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Vuckovic, Study Director — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Stoke Mandevill Hospital, National Spinal Injuries Unit, Stoke Mandeville, Buckinghamshire
  - Queen Elizabeth University Hospital, Queen Elizabeth National Spinal Injurie Unit, Glasgow

IPD SHARING:
Plan to Share IPD: Undecided
Shared on request